CLINICAL TRIAL: NCT04629586
Title: The T1D Exchange Registry
Acronym: T1D Registry
Status: Recruiting | Type: Observational
Sponsor: T1D Exchange, United States (Other)
Responsible Party: Principal Investigator, Kelsie LaFerriere, Lead Research Study Coordinator, T1D Exchange, United States
Other Study IDs: 1822333
Record Dates: First submitted 2020-10-22; First posted 2020-11-16 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-05

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes; Type 1 Diabetes; Diabetes Mellitus
Keywords: insulin; t1d; dm; diabetes; type 1; glucagon
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 50 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals diagnosed with type 1 diabetes: T1D Exchange Registry is currently looking for participants:
  * Of all ages, genders, races, and ethnic groups
  * Living in the United States
  * Diagnosed with type 1 diabetes
  * Currently taking insulin or have had a pancreatic or islet cell transplant
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Observational research study

SUMMARY:
The T1D Exchange Registry is a research study, conducted over time, for individuals with type 1 diabetes and their supporters. Participants volunteer to provide their data for research (for example, by answering questions in annual surveys). Once enrolled, Registry participants have the opportunity to sign up for other studies on various topics related to type 1 diabetes.

To participate, you will be asked to:

* Read and sign an online informed consent form
* Take a survey describing specific demographic and type 1 diabetes management information
* Update your information annually
* Periodically opt in for additional research opportunities (if you choose), i.e. taking new surveys or uploading health device data

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 1 diabetes.
* Individuals younger than 18 years of age must have parent/guardian consent.
* Must be able to read and understand English.
* Currently living in the United States

Exclusion criteria:

* Does not use insulin and has not had a pancreatic or islet cell transplant.
* Cannot fully read and understand English.
* Does not currently live in the United States.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individual diagnosed with type 1 diabetes who can access online Registry.
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2018-12-13 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Gather longitudinal data from individuals living with type 1 diabetes. | 10 years
  Gather longitudinal data on disease, health status, and patient-reported outcomes of individuals living with type 1 diabetes. This will be achieved by presenting participants with annual questionnaires, tracking any changes in their responses over time.

CONTACTS AND LOCATIONS:
Locations (1):
- T1D Exchange, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The information collected in the study may be used in future studies without additional permission from you. This may include research done by other researchers. The information that may be shared will not contain any information that could identify you. There may still be a chance that someone could identify you, but this is not likely. The study results will also be made public. These results will not have any information that could identify you.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code